CLINICAL TRIAL: NCT01403415
Title: A Phase 1 Study of Temsirolimus in Combination With Intensive Re-induction Therapy for Children With Relapsed Acute Lymphoblastic Leukemia and Non-Hodgkin Lymphoma
Brief Title: Temsirolimus, Dexamethasone, Mitoxantrone Hydrochloride, Vincristine Sulfate, and Pegaspargase in Treating Young Patients With Relapsed Acute Lymphoblastic Leukemia or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02679; NCI-2011-02679 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL1114; CDR0000703889; ADVL1114 (Other: COG Phase I Consortium); ADVL1114 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-03

CONDITIONS: Childhood B Acute Lymphoblastic Leukemia; Childhood T Acute Lymphoblastic Leukemia; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Lymphoblastic Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Methotrexate; merphos; Mitoxantrone; pegaspargase; temsirolimus; Sirolimus; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (temsirolimus, combination chemotherapy) (Experimental): Patients receive dexamethasone PO or IV on days 1-5 and 15-19; mitoxantrone hydrochloride IV over 30 minutes on days 1-2; temsirolimus IV over 30 minutes on days 1 and 8; vincristine sulfate IV on days 1, 8, 15, and 22; and pegaspargase IV over 1 hour on days 3 and 17. Some patients may also receive methotrexate IT up to 72 hours prior to or on day 1 and on day 8.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Drug: Pegaspargase; Other: Pharmacological Study; Drug: Temsirolimus; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Other: Pharmacological Study — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase I trial studies the side effects and the best dose of temsirolimus when given together with dexamethasone, mitoxantrone hydrochloride, vincristine sulfate, and pegaspargase in treating young patients with relapsed acute lymphoblastic leukemia or non-Hodgkin lymphoma. Temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, mitoxantrone hydrochloride, vincristine sulfate, and pegaspargase work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving temsirolimus with combination chemotherapy may be and effective treatment for acute lymphoblastic leukemia or non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum-tolerated dose (MTD) and/or recommended phase 2 dose of temsirolimus administered weekly for 2 doses in combination with intensive re-induction chemotherapy in children with relapsed acute lymphoblastic leukemia (ALL) or non-Hodgkin lymphoma (NHL).

II. To define and describe the toxicities of temsirolimus in combination with intensive re-induction chemotherapy in children with relapsed ALL or NHL administered on this schedule.

SECONDARY OBJECTIVES:

I. To compare minimal-residual disease (MRD) levels present at end of induction to historical control in patients with relapsed ALL or NHL with bone marrow involvement of disease.

II. To determine the complete remission (CR) rate in patients with ALL or NHL who receive this regimen.

III. To evaluate responsiveness of patient ALL cells to mammalian target of rapamycin (mTOR) inhibition using in vitro and in vivo pharmacodynamic assessment of the response of ALL blasts to temsirolimus.

OUTLINE: This is a dose-escalation study of temsirolimus.

Patients receive dexamethasone orally (PO) or intravenously (IV) on days 1-5 and 15-19; mitoxantrone hydrochloride IV over 30 minutes on days 1-2; temsirolimus IV over 30 minutes on days 1 and 8; vincristine sulfate IV on days 1, 8, 15, and 22; and pegaspargase IV over 1 hour on days 3 and 17. Some patients may also receive methotrexate intrathecally (IT) up to 72 hours prior to or on day 1 and on day 8.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Patients must have second (2nd) or greater relapse of pre-B ALL, T-cell ALL, lymphoblastic lymphoma, or peripheral T-cell lymphoma; patients may not have refractory disease
  * Patients with leukemia must have had histologic verification of the malignancy at the most recent relapse, including immunophenotyping to confirm diagnosis
* Disease Status:

  * Leukemia: patients with leukemia must have an M3 marrow with or without extramedullary site of relapse OR an M2 bone marrow with an extramedullary site of relapse; patients with central nervous system (CNS) 3 status are not eligible for enrollment
  * Lymphoma: patients with non-Hodgkin lymphoma must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Prior Therapy:

  * Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy, defined as resolution of all such toxicities to =< grade 2 or per the inclusion/exclusion criteria
  * Myelosuppressive chemotherapy:

    * Patients with leukemia or lymphoma who relapse while receiving standard maintenance chemotherapy with steroid, vincristine pulses and oral outpatient chemotherapy will not be required to have a waiting period before enrollment onto this study
    * Patients who relapse while they are not receiving standard maintenance therapy, must have fully recovered from all acute toxic effects of prior therapy; at least 14 days must have elapsed after the completion of cytotoxic therapy, with the exception of hydroxyurea
    * Note: cytoreduction with hydroxyurea in patients can be initiated and continued for up to 24 hours prior to the start of protocol therapy
  * Hematopoietic growth factors: at least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Biologic (anti-neoplastic agent): at least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Immunotherapy: at least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * Monoclonal antibodies: at least 3 half-lives of the antibody after the last dose of a monoclonal antibody with the exception of blinatumomab; patients must have been off blinatumomab infusion for at least 7 days and all drug-related toxicity must have resolved to grade 1 or lower as outline in the inclusion and exclusion criteria
  * Radiation therapy (XRT): at least 14 days after local palliative XRT (small port); at least 84 days must have elapsed if prior total body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial bone marrow (BM) radiation
  * Stem cell infusion: no evidence of active graft versus (vs.) host disease and at least 84 days must have elapsed after transplant or stem cell infusion
  * Study specific limitations on prior therapy: patient may not have received prior therapy with an mTOR inhibitor
  * Note: intrathecal (IT) methotrexate (MTX) that is given up to 72 hours prior to initiation of systemic chemotherapy per ADVL1114 counts as protocol therapy and not prior anti-cancer therapy; IT MTX given > 72 hours prior does not count as protocol therapy
* Platelet count >= 20,000/mm^3 (may receive platelet transfusions) to initiate therapy

  * Patients must not be known to be refractory to red cell or platelet transfusion
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 225 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Gamma-glutamyl transpeptidase (GGT) =< ULN for age
* Serum albumin >= 2 g/dL
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study
* Pulse oximetry > 94% on room air
* Baseline chest x-ray; patients with active infectious disease or pneumonitis are not eligible
* Serum triglyceride level =< 300 mg/dL and serum cholesterol level =< 300 mg/dL
* Random or fasting blood glucose within the upper normal limits for age; if the initial blood glucose is a random sample that is above the upper normal limits, then a follow-up fasting blood glucose can be obtained and must be within the upper normal limits for age
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients receiving stable or decreasing doses of corticosteroids for =< 7 days prior to enrollment, or who are receiving increasing doses of corticosteroids, are not eligible for enrollment; the exception to this is pulsed steroids used for maintenance chemotherapy
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible (except patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy)
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who cannot receive asparaginase are not permitted on trial; substitution with Asparaginase Erwinia Chrysanthemi is acceptable
* Cumulative prior anthracycline exposure must not exceed 400 mg/m^2 (each 10 mg/m^2 of idarubicin or mitoxantrone should be calculated as the isotoxic equivalent of 30 mg/m^2 of daunorubicin or doxorubicin)
* Patients who are currently receiving therapeutic anticoagulants (including aspirin, low molecular weight heparin, and others) are not eligible
* Patients who are currently receiving angiotensin-converting enzyme (ACE) inhibitors are not eligible due to the development of angioneurotic edema-type reactions in some subjects who received concurrent treatment with temsirolimus + ACE inhibitors
* Enzyme-Inducing anti-convulsants: patients who are currently receiving enzyme-inducing anti-convulsants (i.e., phenytoin, phenobarbital, or carbamazepine) are not eligible
* Patients with CNS 3 status at enrollment are not eligible
* Patients must have no pre-existing grade 1 or higher ulcerations, fistulas, mucosal lesions, or skin barrier breakdown
* Patients who have an uncontrolled infection are not eligible
* Patients with known optic nerve and/or retinal involvement (because it may not be possible to safely delay irradiation) are not eligible; patients presenting with visual disturbances by history or physical exam should have an ophthalmological exam and magnetic resonance imaging (MRI) within 14 days prior to enrollment to determine whether there is optic nerve or retinal involvement
* Patients with known Down syndrome, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of temsirolimus in combination with intensive re-induction chemotherapy graded according to the NCI CTCAE v4.0 | Up to 30 days post-treatment
  A descriptive summary of all toxicities will be reported.
MTD and/or recommended phase II dose defined as the maximum dose at which fewer than one-third of patients experience dose-limiting toxicity graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to day 36
  A descriptive summary of all toxicities will be reported.

SECONDARY OUTCOMES:
CR rate according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 30 days post-treatment
MRD levels present at the end of induction | Up to 30 days post-treatment
  Compared to a historical control in patients with bone marrow involvement of disease using a t-test or nonparametric analog.
mTOR inhibitor effects on downstream signaling in patient lymphoblasts In vitro and in vivo | Up to 30 days post-treatment
  The pharmacodynamic data will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rheingold, Principal Investigator — COG Phase I Consortium
Locations (31):
- United States (30):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada